CLINICAL TRIAL: NCT06250933
Title: The Effect of Nursing Approach Grounded in Meleis's Transition Theory on Postpartum Depression, Maternal Self-Efficacy, and Breastfeeding Self-Efficacy in Women Experiencing Preterm Birth
Brief Title: The Meleis Theory on Postpartum Depression, Breastfeeding, and Maternal Self-Efficacy in Women Experiencing Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Rahime Aksoy, Research Assistant, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SBU-AKSOYGUVENC1
Record Dates: First submitted 2024-01-08; First posted 2024-02-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-02

CONDITIONS: Premature Birth; Theory, Double Bind; Postpartum Depression; Breast Feeding; Self Efficacy
Keywords: premature birth; Theory; Postpartum Depression; Breastfeeding; Self efficacy
MeSH Terms: conditions — Premature Birth; Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Following recruitment, the women were divided into a study and a control group by randomization (1:2 randomization)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment group (Experimental): In the intervention group, training and counseling were provided within the scope of the nursing approach based on Meleis transition theory. In this context, training consisting of three sessions of 100 minutes in total was given and counseling was provided by conducting 3-4 interviews by phone in the following weeks. In the interviews, counseling was provided on the issues that women needed, especially the difficulties they faced in the postpartum period, postpartum depression symptoms, self-care, breastfeeding problems and maternal self-efficacy. In this process, the women were evaluated three times in total, in the first postpartum week (pre-test), two weeks after delivery (post-test 1) and 42nd day (6th week) (post-test 2) with the Breastfeeding Self-Efficacy Scale, Perceived Maternal Self-Efficacy Scale and Edinburgh Postpartum Depression Scale.
  Translated with DeepL.com (free version)
  Interventions: Other: Postpartum Maternal Care and Premature Infant Care Training
- Control group (No Intervention): The control group will continue to receive routine care

INTERVENTIONS:
Other: Postpartum Maternal Care and Premature Infant Care Training — Training and counseling were provided. In this context, training consisting of three sessions of 100 minutes in total was provided and counseling was provided in the following weeks by conducting 3-4 telephone interviews.
  The intervention involves the provision of a training and counseling program designed to increase women's breastfeeding and maternal self-efficacy and reduce the risk of postpartum depression.
  In the training phase, women will receive training on postpartum maternal care and premature infant care.
  Arms: Experiment group

SUMMARY:
The aim of this study was to evaluate the effect of a nursing approach based on Meleis' Transition Theory on postpartum depression, maternal self-efficacy and breastfeeding self-efficacy in women who gave birth preterm. The randomized controlled study was conducted in the Neonatal Intensive Care Unit. The study sample consisted of preterm women who volunteered to participate in the study and met the inclusion criteria. A training guide was prepared within the scope of the nursing approach based on Transition Theory. After the theoretical training in the second week after delivery, the intervention group received counseling through face-to-face and telephone individual interviews, while the control group received routine care only in the hospital. Scales were administered to women in both groups at the first interview, 2 weeks later and on day 42.

DETAILED DESCRIPTION:
The study will be conducted in the Maternity Hospital and Level 3 Neonatal Intensive Care Unit (NICU) of a hospital in Turkey. Ethical principles were taken into consideration in the study. After the necessary arrangements were made in the data collection forms, the participants were given written and verbal explanations about the study and their informed consent was obtained. Data collection forms were applied individually through face-to-face interviews with women who volunteered to participate in the study. training and counseling were provided within the scope of nursing approach. In this context, training consisting of three sessions of 100 minutes in total was given and counseling was provided in the following weeks by conducting 3-4 interviews by phone. In the interviews, counseling was provided on the issues that women needed, especially the difficulties they faced in the postpartum period, postpartum depression symptoms, self-care, breastfeeding problems and maternal self-efficacy. During this period, the women were evaluated with the Breastfeeding Self-Efficacy Scale, the Perceived Maternal Self-Efficacy Scale and the Edinburgh Postnatal Depression Scale three times in total: the first week postpartum (pre-test), two weeks postpartum (post-test 1) and 42 days (week 6) (post-test 2). No intervention other than routine hospital practices was performed on these women. Personal data form, Breastfeeding Self-Efficacy Scale, Perceived Maternal Self-Efficacy Scale, and Edinburgh Postpartum Depression Scale were administered at initial admission. Two weeks after birth and on day 42, the Breastfeeding Self-Efficacy Scale, Perceived Maternal Self-Efficacy Scale and Edinburgh Postpartum Depression Scale were administered again, and then a training booklet on the nursing approach based on the Meleis Transition Theory was given.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Without communication barriers
* Literate
* Married
* Not undergoing psychological treatment
* Preterm birth occurring between gestational weeks 28-32
* Mothers of preterm infants receiving continuous treatment in the NICU (Neonatal Intensive Care Unit) at the time of data collection
* Not having received breastfeeding education from healthcare professionals

Exclusion Criteria:

* The baby dies during the treatment process
* Not participating in the stages of the research
* Asking to withdraw from the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Postpartum Depression | The first week postpartum
  The Edinburgh Postnatal Depression Scale (EPDS), developed by Cox et al. (1987), is a screening tool designed to assess the risk of depression in women during the postnatal period. It is not intended for the diagnosis of depression. The EPDS is a self-report scale consisting of 10 items, rated on a 4-point Likert scale. Responses with four options are scored between 0 and 3, with the lowest possible score being 0 and the highest 30. In the assessment, items 1, 2, and 4 are scored as 0, 1, 2, 3, while items 3, 5, 6, 7, 8, 9, and 10 are scored in reverse as 3, 2, 1, 0.The cutoff point for the EPDS was calculated as 13, and women with scores of 13 or higher were considered at risk.
Maternal Self-Efficacy | The first week postpartum
  The Perceived Maternal Self-Efficacy Scale This scale was developed by Barnes and Adamson-Macedo (2007) and its Turkish validity and reliability were examined by Kadiroğlu (2018). The scale assesses the perceived maternal self-efficacy levels of mothers with prematurely born infants hospitalized in a neonatal intensive care unit. The reliability coefficient for mothers of prematurely born infants in the hospital is 0.98. The scale, consisting of 19 items, is rated on a 1 to 4 scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree). Scores obtained are summed to calculate the scale score, ranging from 19 to 76. A higher score indicates a higher perceived maternal self-efficacy level.
Breastfeeding Self-Efficacy | The first week postpartum
  Breastfeeding Self-Efficacy Scale for Mothers of Preterm Infants Developed by Wheeler & Dennis (2013), this scale is based on the 14-item 'Breastfeeding Self-Efficacy Scale-Short Form' developed by Dennis (2003) and has undergone Turkish reliability and validity testing by Aluş Tokat et al. (2020). Four additional items related to the breastfeeding of hospitalized and/or preterm infants were included. The resulting modified scale comprises 18 items. The scale, utilized among English-speaking Canadian mothers with hospitalized or premature infants, demonstrated a Cronbach's alpha internal consistency of 0.88 (Wheeler and Dennis, 2013). The scale is a 5-point Likert Type scale, where 1= "Not at all confident" and 5= "Always confident." All items are positively phrased. The minimum and maximum scores that can be obtained from the scale are 18 and 90, respectively. A higher score indicates a higher level of breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Postpartum Depression | Two weeks postpartum
  The Edinburgh Postnatal Depression Scale (EPDS), developed by Cox et al. (1987), is a
Maternal Self-Efficacy | Two weeks postpartum
  The Perceived Maternal Self-Efficacy Scale This scale was developed by Barnes and Adamson-Macedo (2007) and its Turkish validity and reliability were examined by Kadiroğlu (2018). The scale assesses the perceived maternal self-efficacy levels of mothers with prematurely born infants hospitalized in a neonatal intensive care unit. The reliability coefficient for mothers of prematurely born infants in the hospital is 0.98. The scale, consisting of 19 items, is rated on a 1 to 4 scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree). Scores obtained are summed to calculate the scale score, ranging from 19 to 76. A higher score indicates a higher perceived maternal self-efficacy level.
Breastfeeding Self-Efficacy | Two weeks postpartum
  Breastfeeding Self-Efficacy Scale for Mothers of Preterm Infants Developed by Wheeler & Dennis (2013), this scale is based on the 14-item 'Breastfeeding Self-Efficacy Scale-Short Form' developed by Dennis (2003) and has undergone Turkish reliability and validity testing by Aluş Tokat et al. (2020). Four additional items related to the breastfeeding of hospitalized and/or preterm infants were included. The resulting modified scale comprises 18 items. The scale, utilized among English-speaking Canadian mothers with hospitalized or premature infants, demonstrated a Cronbach's alpha internal consistency of 0.88 (Wheeler and Dennis, 2013). The scale is a 5-point Likert Type scale, where 1= "Not at all confident" and 5= "Always confident." All items are positively phrased. The minimum and maximum scores that can be obtained from the scale are 18 and 90, respectively. A higher score indicates a higher level of breastfeeding self-efficacy.

OTHER OUTCOMES:
Postpartum Depression | On the 42nd day postpartum
  The Edinburgh Postnatal Depression Scale (EPDS), developed by Cox et al. (1987), is a screening tool designed to assess the risk of depression in women during the postnatal period. It is not intended for the diagnosis of depression. The EPDS is a self-report scale consisting of 10 items, rated on a 4-point Likert scale. Responses with four options are scored between 0 and 3, with the lowest possible score being 0 and the highest 30. In the assessment, items 1, 2, and 4 are scored as 0, 1, 2, 3, while items 3, 5, 6, 7, 8, 9, and 10 are scored in reverse as 3, 2, 1, 0.The cutoff point for the EPDS was calculated as 13, and women with scores of 13 or higher were considered at risk.
Maternal Self-Efficacy | On the 42nd day postpartum
  The Perceived Maternal Self-Efficacy Scale This scale was developed by Barnes and Adamson-Macedo (2007) and its Turkish validity and reliability were examined by Kadiroğlu (2018). The scale assesses the perceived maternal self-efficacy levels of mothers with prematurely born infants hospitalized in a neonatal intensive care unit. The reliability coefficient for mothers of prematurely born infants in the hospital is 0.98. The scale, consisting of 19 items, is rated on a 1 to 4 scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree). Scores obtained are summed to calculate the scale score, ranging from 19 to 76. A higher score indicates a higher perceived maternal self-efficacy level.
Breastfeeding Self-Efficacy | On the 42nd day postpartum
  Breastfeeding Self-Efficacy Scale for Mothers of Preterm Infants Developed by Wheeler & Dennis (2013), this scale is based on the 14-item 'Breastfeeding Self-Efficacy Scale-Short Form' developed by Dennis (2003) and has undergone Turkish reliability and validity testing by Aluş Tokat et al. (2020). Four additional items related to the breastfeeding of hospitalized and/or preterm infants were included. The resulting modified scale comprises 18 items. The scale, utilized among English-speaking Canadian mothers with hospitalized or premature infants, demonstrated a Cronbach's alpha internal consistency of 0.88 (Wheeler and Dennis, 2013). The scale is a 5-point Likert Type scale, where 1= "Not at all confident" and 5= "Always confident." All items are positively phrased. The minimum and maximum scores that can be obtained from the scale are 18 and 90, respectively. A higher score indicates a higher level of breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Rahime AKSOY BULGURCU, Principal Investigator — Bilecik Seyh Edebali Universitesi
Locations (1):
- Rahime AKSOY BULGURCU, Bilecik, Gülümbe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No